CLINICAL TRIAL: NCT01562756
Title: Pilot for Patient Response to Spinal Manipulation (PRiSM)
Brief Title: Patient Response to Spinal Manipulation - Pilot Study
Acronym: PRiSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRiSM Pilot; U19AT004663 (NIH)
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HVLA-SM (Experimental): High velocity, low amplitude lumbo-pelvic manipulation
  Interventions: Other: HVLA-SM

INTERVENTIONS:
Other: HVLA-SM — High velocity, low amplitude spinal manipulation

SUMMARY:
In collaboration with the University of Iowa, the Palmer Center for Chiropractic Research will conduct a pilot study for the purposes of testing equipment, finalizing data collection protocol, and training study personnel before conducting the full-scale trial.

DETAILED DESCRIPTION:
In collaboration with the University of Iowa, the Palmer Center for Chiropractic Research will conduct a pilot study for the purposes of testing equipment, finalizing the data collection protocol, and training study personnel before conducting the full-scale trial. Only feasibility data will be collected and reported for this pilot study.

The full-scale trial, titled as "Patient response to spinal manipulation" (Trial registration: NCT01670292 on clinicaltrials.gov), is the Project 1 of the Developmental Center for Clinical and Translational Science in Chiropractic (Award No. U19AT004663).

In the current pilot study, we test how research clinicians can treat patients under study measurement conditions and with equipment resulting in modified treatment procedures. This pilot study will also test spinal stiffness using 3 different methods on 2 study visits. We will also assess the function of low back muscles during standing and while bending forward on 2 visits. These measurements include placing sensors on the back with tape and measuring the electrical activity of low back muscles. Participants with low back pain are treated with side-lying high-velocity low-amplitude spinal manipulation by experienced research clinicians who are doctors of chiropractic. Specifically, we will recruit 6 participants who are 21 - 64 years old and have had low back pain for at least 3 months. Each participant will attend 1 baseline visit, 1 enrollment visit, and 4 treatment visits over a period of approximately 4 weeks. Following the baseline visit, participant eligibility will be determined. The enrollment visit will be scheduled on the same day as the first treatment visit. The following feasibility data will be collected:

* # of participants recruited
* # of participants consented
* # of participants enrolled
* # of participants who completed the study
* Total duration of the study from launch data to the final study visit

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* Signed informed consent document
* Chronic (12+ weeks) low back pain (LBP)
* Average pain within past 24 hours ≥ 2/10 at phone screen, baseline visit 1, and baseline visit 2

Exclusion Criteria:

* Compliance concerns such as refusal to shave body hair
* No manipulable lesion in L3, L4, L5 or SI joints (The absence of typical palpatory characteristics as well as the absence of a global assessment that would indicate that spinal manipulation is likely to generate a positive therapeutic effect, even without the presence of standard palpatory findings)
* Comorbid Conditions:
* Serious Contaminant Illness
* Inflammatory or Destructive Spinal Tissue change
* Ankylosing Spondylitis
* Fibromyalgia
* Rheumatoid Arthritis
* Neuromuscular Disease (e.g. Parkinson's, Muscular Dystrophy, Cerebral Palsy, or Myasthenia gravis)
* Spinal Surgery < 6 mo
* Suspicion of drug or alcohol abuse
* Uncontrolled hypertension
* Peripheral Arterial Disease
* Undetermined, infectious or visceral source of LBP
* Other comorbid conditions prohibiting treatment and/or testing
* Safety Concerns
* Bleeding Disorders
* Contraindications to HVLA-SM
* Quebec Task Force (QTF) criterion 4-11:
* QTF 4: Pain + radiation to upper/lower limb with signs
* QTF 5: Presumptive compression of a spinal nerve root on a simple roentgenogram
* QTF 6: Compression of a spinal nerve root confirmed by specific imaging techniques
* QTF 7: Spinal Stenosis
* QTF 8: Postsurgical status, 1-6 months after intervention
* QTF 9: Postsurgical status, >6 months after intervention
* QTF 10: Chronic pain syndrome
* QTF 11: Other diagnoses
* Pregnancy
* Pacemaker or defibrillator
* Inability to read or verbally comprehend English
* Joint Replacement
* Sensitivity to adhesive
* Additional diagnostic procedures other than x-ray necessary
* BDI-II > 29
* Retention of legal advice and open or pending case related to LBP
* BMI > 40
* Unwilling to have low back and wrist shaved
* Seeking or receiving compensation for any disability?

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ting Xia, PhD, Principal Investigator — Palmer College of Chiropractic
Locations (1):
- Palmer College of Chiropractic, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Feasibility/pilot study

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HVLA-SM
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HVLA-SM
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Conducting a Full-scale Randomized Control Trial to Evaluate Patient Response to Spinal Manipulation: Number of Participants Who Were Recruited, Consented, Enrolled, and Completed the Study
Description: Feasibility was measured by the numbers of participants: recruited, consented, enrolled, and retained. This pilot study allowed for testing of equipment, finalizing the data collection protocol, and training study personnel before conducting the full-scale trial.
Time Frame: Approximately 4-6 weeks including initial eligibility screening, baseline visits, and 2 weeks of treatment visits
Measure: Number; unit: participants
Groups:
- Feasibility Outcomes: The feasibility outcomes (Primary outcomes 1 & 2) for this study include participant recruitment, enrollment, and the duration of the study.
Arm/Group | Feasibility Outcomes
Number analyzed (Participants) | 6
participants
  # Participants Recruited | 19
  # Participants Consented | 9
  # Participants Enrolled | 6
  # Participants Completed | 6

2. Primary Outcome: Feasibility of Conducting a Full-scale Randomized Control Trial to Evaluate Patient Response to Spinal Manipulation: Study Duration.
Description: Feasibility was measured by the study duration from study launch to collection of final study outcomes. This pilot study allowed for testing of equipment, finalizing the data collection protocol, and training study personnel before conducting the full-scale trial.
Time Frame: Approximately 4-6 weeks including initial eligibility screening, baseline visits, and 2 weeks of treatment visits
Measure: Number; unit: months
Units Other Than Participants: months
Arm/Group | Feasibility Outcomes
Number analyzed (Participants) | 6
Number analyzed (months) | 4
months | 4

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | HVLA-SM
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes